CLINICAL TRIAL: NCT05298722
Title: Prediction of Surgical Resectability After FOLFIRINOX Chemotherapy for Borderline Resectable and Locally Advanced Pancreatic Cancer: the Role of Diffusion Weighted Magnetic Resonance Imaging, Radiomics and Liquid Biopsy
Brief Title: Prediction of Surgical Resectability After FOLFIRINOX Chemotherapy for Borderline Resectable and Locally Advanced Pancreatic Cancer: the Role of Diffusion Weighted Magnetic Resonance Imaging, Radiomics and Liquid Biopsy (PeRFormanCe Trial)
Acronym: PeRFormanCe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ONZ-2022-0088 - PeRFormanCe
Record Dates: First submitted 2021-11-22; First posted 2022-03-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Magnetic Resonance Imaging; Radiomics; Liquid Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study arm (Other): Imaging with CT-scan and MRI-DWI and peripheral blood samples for liquid biopsy
  Interventions: Diagnostic Test: Imaging analysis of CT-scan and MRI with radiomics and genetic analysis of peripheral blood samples and questionnaires.

INTERVENTIONS:
Diagnostic Test: Imaging analysis of CT-scan and MRI with radiomics and genetic analysis of peripheral blood samples and questionnaires. — * The images from CT scans and MRI with DWI will be processed using specialized software to determine the direction of diffusion tensors. This will indicate the diffusion direction using color coding (red, green, and blue for the x, y, and z components of the vector) and the intensity using anisotropy (brightness of voxels). Further analysis will be performed using fiber tracking, which provides a clear representation of the functional connectivity of adjacent tissues.
  * Genetic profiling of liquid biopsies: Multi-omics profiling of liquid biopsies (blood samples) will be conducted, followed by cell phenotyping, longitudinal analysis of driver mutations and epigenetic changes in cfDNA, and genotyping of germline variations.
  * Questionnaires for patient-reported outcomes and health economic analysis:
  EQ-5D-5L PAN 26 HADS
  Other Names: Analysis of imaging with radiomics and genetic analysis of peripheral blood samples (liquid biopsy)

SUMMARY:
In this prospective study, new diagnostic tools will be explored for patients with borderline resectable and locally advanced pancreatic ductal adenocarcinoma (BR or LAPDA) who undergo neoadjuvant chemotherapy with FOLFIRINOX. The diagnostic work-up and therapy for the study population will not differ from the gold standard during the study; only additional diagnostic tools will be implemented, and their value will be analyzed post hoc.

The 5-year survival rate of pancreatic cancer is 9%, but this can be drastically improved if surgery is possible. With its increasing incidence and poor prognosis, pancreatic cancer is becoming a global oncologic challenge where major breakthroughs are still required to improve patient outcomes. Patients with BR or LAPDA typically undergo neoadjuvant treatment with FOLFIRINOX chemotherapy, followed by referral for surgery if a response is observed. In these cases, surgical resectability is difficult to predict based on CT imaging due to the tumor's desmoplastic reaction, which obscures tumor-vessel contact without clear morphological changes. Consequently, patients without tumor progression on CT and with a decreased tumor marker (CA 19-9) are considered for surgical exploration to ensure that no potentially curative treatment is denied. However, the non-specific nature of CA 19-9 and the unreliable spatial changes on CT do not allow for accurate patient stratification. Therefore, alternative diagnostic strategies are needed to better predict resectability, minimizing unnecessary laparotomies while ensuring that potentially curative approaches are not overlooked.

In this project, the investigator will apply diffusion-weighted magnetic resonance imaging (DW-MRI), as it has been shown to be useful in assessing tumor response beyond morphological parameters. DW-MRI enables the detection of functional tumor changes, variations in vascularization, and fibrosis without modifications in shape. The statistical evaluation of visual information using radiomics optimizes data analysis, allowing comparisons over time (before and after chemotherapy) and correlation with operative findings (resectable or unresectable tumor).

The investigator will focus on patients with BR and LAPDA and assess whether a combination of clinical and genetic factors can predict successful surgical resection. To this end, DW-MRI imaging will be complemented by multi-omics profiling in liquid biopsies. Furthermore, the investigator aims to validate, in a prospective patient cohort, the predictive value of recently published single nucleotide polymorphisms (SNPs) in genes that regulate cancer progression, invasion, and metastasis. Some alleles of these SNPs have been associated with an increased risk of tumor-related mortality compared to protective genotypes.

DETAILED DESCRIPTION:
Study Aim The aim of this study is to assess whether the combination of radiomics, diffusion-weighted magnetic resonance imaging (DW-MRI), and multi-omics profiling in liquid biopsies-both before and after neoadjuvant chemotherapy-can predict the probability of achieving successful surgical excision in patients with borderline resectable (BR) and locally advanced pancreatic ductal adenocarcinoma (LAPDA).

Additionally, a subgroup analysis will be performed, taking into account risk alleles of single nucleotide polymorphisms (SNPs) that have recently been associated with worse survival outcomes.

The primary endpoint of this study is to improve the prediction of surgical resectability following neoadjuvant chemotherapy with FOLFIRINOX in patients with BR and LAPDA. The focus is on increasing diagnostic specificity to better identify patients with unresectable tumors, thereby avoiding unnecessary exploratory laparotomies that may delay further chemotherapy.

Secondary endpoints include the evaluation of postoperative complications, cost minimization, and disease-free and overall survival.

Background & Rationale All factors evaluated in this study-DW-MRI, radiomics, genetic markers (SNPs), and multi-omics profiling in liquid biopsies-have individually shown promise for early diagnosis, prognosis assessment, and correlation with tumor response to chemotherapy in pancreatic cancer. However, these modalities have never been combined in an innovative study such as this, where they are integrated to enhance clinical decision-making.

This project aims to apply existing knowledge to have an immediate impact on therapeutic decision-making, reducing unnecessary surgical explorations and ultimately improving patient quality of life while optimizing treatment efficiency.

Patients with BR or LAPDA typically undergo neoadjuvant treatment with FOLFIRINOX, followed by referral for surgery if they respond to chemotherapy. However, surgical resectability is challenging to predict using CT imaging alone, as the tumor's desmoplastic reaction can obscure tumor-vessel contact without clear morphological changes. As a result, patients with stable disease on CT and a decreased CA 19-9 level are considered for surgical exploration to ensure that no potentially curative treatment is withheld.

Since CA 19-9 is non-specific and CT lacks reliable spatial resolution for detecting subtle tumor changes, alternative strategies are needed to improve resectability predictions and avoid negative laparotomies. DW-MRI has demonstrated its value in evaluating tumor response beyond morphological parameters, while radiomics can enhance data analysis. Additionally, multi-omics profiling using liquid biopsies has shown a correlation with tumor response to chemotherapy in pancreatic cancer, though its utility in the neoadjuvant setting remains unclear.

Objective This multicenter prospective study aims to assess the utility of DW-MRI, radiomics, and liquid biopsy in predicting tumor resectability after neoadjuvant treatment with FOLFIRINOX in patients with BR and LAPDA.

When chemotherapy results in a reduction of CA 19-9 but no significant morphological change on CT, some tumors may still be eligible for an R0 resection. The investigator hypothesizes that these cases can be preoperatively identified by detecting a reduction in multi-omics markers in liquid biopsies, along with decreased vascularity and cellularity in the tumor-vessel interface on DW-MRI.

Study Design A prospective interventional study with a single study arm.

Study Population Patients with BR or LAPDA scheduled for neoadjuvant chemotherapy with FOLFIRINOX and without contraindications for pancreatic surgery.

A minimum sample size of 45 patients undergoing surgical exploration has been calculated (80% power, α = 0.05, two-tailed).

Intervention Patients with BR and LAPDA will be discussed in a multidisciplinary oncologic meeting and will receive standard-of-care treatment. In addition to routine clinical evaluation, CT imaging, and CA 19-9 assessment before and after chemotherapy, participants will undergo DW-MRI and provide a peripheral blood sample for multi-omics profiling in liquid biopsies.

If no tumor progression is observed on imaging and CA 19-9 levels decrease post-chemotherapy, patients will be considered for surgical exploration. During surgery, a blood sample will be collected from the supra-pancreatic portal vein to measure circulating tumor cells (CTCs) before and after tumor resection-if an R0 resection is feasible.

Additionally, a peripheral blood sample will be taken at the first postoperative consultation to analyze multi-omics profiling in liquid biopsies and CA 19-9 levels.

Burden, Risks, and Benefits of Participation Compared to standard care, participants in this study will undergo two additional DW-MRI scans and provide extra peripheral blood samples.

DW-MRI is a widely used, safe imaging modality, and blood samples are routinely collected as part of oncologic treatment. The study aims to refine surgical decision-making, minimizing unnecessary procedures and ultimately improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, aged 18 years and above
* Diagnosis of BR or LA PDAC according to NCCN guidelines (version 1.2020)
* Histologic diagnosis of PDAC
* No medical or anesthetic contra-indication for surgery
* Able to understand nature of the study procedures
* Willing to participate and give written informed consent

Exclusion Criteria:

* Age < 18 years
* Distant metastases
* Histologic diagnosis of cholangiocarcinoma, duodenal carcinoma or neuroendocrine tumor
* Known hypersensitivity for MRI contrast
* Pacemaker or prosthesis with incompatibility for MRI
* Claustrophobia
* Pregnancy or breastfeeding
* Not able to understand nature of the study procedure
* Performance status ECOG score: >2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Prediction of surgical resectability | 2 years
  Create an algorithm to predict surgical resectability of BR and LA PDAC after neoadjuvant FOLFIRINOX with radiomics analysis of CT and DW-MRI to determine the tumoral vascular invasion in combination with the evolution of CA19-9 and genetic profilling of liquid biopsies (phenotyping and quantification of the CTCs, longitudinal analysis of driver mutations and epigenetic changes in cfDNA).
R1 resection rate | 2 years
Histopathological response | 2 years

SECONDARY OUTCOMES:
Prediction of R0 resection | 2 years
  Create an algorithm to predict R0 surgical resectability of BR and LA PDAC after neoadjuvant FOLFIRINOX with radiomics analysis of CT and DW-MRI to determine the tumoral vascular invasion in combination with the evolution of CA19-9 and genetic profilling of liquid biopsies (phenotyping and quantification of the CTCs, longitudinal analysis of driver mutations and epigenetic changes in cfDNA).
Perioperative complications | 2 years
  Evaluation according to Clavien-Dindo classification
Generic measurement of health status | 4 years
  Questionnaire EQ-5D-5L
Overall survival | 4 years
Disease free survival | 4 years
Measurement of quality of life in patients with pancreatic cancer | 4 years
  Questionnaire PAN 26

CONTACTS AND LOCATIONS:
Locations (8):
- Belgium (7):
  - Ghent University Hospital, Ghent, East Flanders
  - AZ Sint Blasius Dendermonde, Dendermonde
  - AZ Alma Eeklo, Eeklo
  - AZ Jan Palfijn Ghent, Ghent
  - AZ Sint Lucs Ghent, Ghent
  - AZ Oudenaarde, Oudenaarde
  - AZ Vitaz Sint Niklaas - Lokeren, Sint-Niklaas
- ZorgSaam ZH DeHonte Terneuzen, Terneuzen, Zeeland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
If a multicentric study should arise in the future to combine data of this subpopuplation of patients with pancreatic cancer, it would be interesting to analyze a larger studypopulation in order to possibly achieve more signicant conclusions.

REFERENCES:
- [Background] Isaji S, Mizuno S, Windsor JA, Bassi C, Fernandez-Del Castillo C, Hackert T, Hayasaki A, Katz MHG, Kim SW, Kishiwada M, Kitagawa H, Michalski CW, Wolfgang CL. International consensus on definition and criteria of borderline resectable pancreatic ductal adenocarcinoma 2017. Pancreatology. 2018 Jan;18(1):2-11. doi: 10.1016/j.pan.2017.11.011. Epub 2017 Nov 22. PMID 29191513
- [Background] Marchegiani G, Todaro V, Boninsegna E, Negrelli R, Sureka B, Bonamini D, Salvia R, Manfredi R, Pozzi Mucelli R, Bassi C. Surgery after FOLFIRINOX treatment for locally advanced and borderline resectable pancreatic cancer: increase in tumour attenuation on CT correlates with R0 resection. Eur Radiol. 2018 Oct;28(10):4265-4273. doi: 10.1007/s00330-018-5410-6. Epub 2018 Apr 20. PMID 29679211
- [Background] Gemenetzis G, Groot VP, Yu J, Ding D, Teinor JA, Javed AA, Wood LD, Burkhart RA, Cameron JL, Makary MA, Weiss MJ, He J, Wolfgang CL. Circulating Tumor Cells Dynamics in Pancreatic Adenocarcinoma Correlate With Disease Status: Results of the Prospective CLUSTER Study. Ann Surg. 2018 Sep;268(3):408-420. doi: 10.1097/SLA.0000000000002925. PMID 30080739
- [Background] Tang L, Zhou XJ. Diffusion MRI of cancer: From low to high b-values. J Magn Reson Imaging. 2019 Jan;49(1):23-40. doi: 10.1002/jmri.26293. Epub 2018 Oct 12. PMID 30311988
- [Background] Rebelo et al. Circulating tumor cells in pancreatic cancer: a review. Journal of pancreatology (2019) 2:2.
- [Background] Dimitrakopoulos C, Vrugt B, Flury R, Schraml P, Knippschild U, Wild P, Hoerstrup S, Henne-Bruns D, Wuerl P, Graf R, Breitenstein S, Bond G, Beerenwinkel N, Grochola LF. Identification and Validation of a Biomarker Signature in Patients With Resectable Pancreatic Cancer via Genome-Wide Screening for Functional Genetic Variants. JAMA Surg. 2019 Jun 1;154(6):e190484. doi: 10.1001/jamasurg.2019.0484. Epub 2019 Jun 19. PMID 30942874
- [Background] Okubo K, Uenosono Y, Arigami T, Mataki Y, Matsushita D, Yanagita S, Kurahara H, Sakoda M, Kijima Y, Maemura K, Natsugoe S. Clinical impact of circulating tumor cells and therapy response in pancreatic cancer. Eur J Surg Oncol. 2017 Jun;43(6):1050-1055. doi: 10.1016/j.ejso.2017.01.241. Epub 2017 Feb 12. PMID 28233633
- [Background] Poruk KE, Valero V 3rd, Saunders T, Blackford AL, Griffin JF, Poling J, Hruban RH, Anders RA, Herman J, Zheng L, Rasheed ZA, Laheru DA, Ahuja N, Weiss MJ, Cameron JL, Goggins M, Iacobuzio-Donahue CA, Wood LD, Wolfgang CL. Circulating Tumor Cell Phenotype Predicts Recurrence and Survival in Pancreatic Adenocarcinoma. Ann Surg. 2016 Dec;264(6):1073-1081. doi: 10.1097/SLA.0000000000001600. PMID 26756760
- [Background] Poruk KE, Blackford AL, Weiss MJ, Cameron JL, He J, Goggins M, Rasheed ZA, Wolfgang CL, Wood LD. Circulating Tumor Cells Expressing Markers of Tumor-Initiating Cells Predict Poor Survival and Cancer Recurrence in Patients with Pancreatic Ductal Adenocarcinoma. Clin Cancer Res. 2017 Jun 1;23(11):2681-2690. doi: 10.1158/1078-0432.CCR-16-1467. Epub 2016 Oct 27. PMID 27789528
- [Background] Harouaka RA, Nisic M, Zheng SY. Circulating tumor cell enrichment based on physical properties. J Lab Autom. 2013 Dec;18(6):455-68. doi: 10.1177/2211068213494391. Epub 2013 Jul 5. PMID 23832928
- [Background] Sollier E, Go DE, Che J, Gossett DR, O'Byrne S, Weaver WM, Kummer N, Rettig M, Goldman J, Nickols N, McCloskey S, Kulkarni RP, Di Carlo D. Size-selective collection of circulating tumor cells using Vortex technology. Lab Chip. 2014 Jan 7;14(1):63-77. doi: 10.1039/c3lc50689d. Epub 2013 Sep 23. PMID 24061411
- [Background] Kolostova K, Rzechonek A, Schutzner J, Grill R, Lischke R, Hladik P, Simonek J, Bobek V. Circulating Tumor Cells as an Auxiliary Diagnostic Tool in Surgery. In Vivo. 2017 Nov-Dec;31(6):1197-1202. doi: 10.21873/invivo.11190. PMID 29102946
- [Background] Bobek V, Gurlich R, Eliasova P, Kolostova K. Circulating tumor cells in pancreatic cancer patients: enrichment and cultivation. World J Gastroenterol. 2014 Dec 7;20(45):17163-70. doi: 10.3748/wjg.v20.i45.17163. PMID 25493031
- [Derived] Abreu de Carvalho LF, Gryspeerdt F, Ceelen W, Geboes K, Ribeiro S, Hoorens A, Vandenbussche N, Claes KBM, Lecluyse C, Anisau A, Van Ongeval J, Lybaert W, Triest L, Vervaecke A, Sas S, Claerhout B, Beyls C, Sie M, Berrevoet F. Prediction of surgical resectability after FOLFIRINOX chemotherapy for borderline resectable and locally advanced pancreatic cancer (PeRFormanCe): a multicenter prospective trial - trial protocol. BMC Surg. 2025 May 13;25(1):204. doi: 10.1186/s12893-025-02938-1. PMID 40361171